CLINICAL TRIAL: NCT02264743
Title: Comparison of Ultra-low-dose Oral Versus Trans-dermal Hormone Therapy on Coagulation Activation and Metabolic Risk Factors for Cardiovascular Disease
Brief Title: Oral Verses Patch Trial In Menopausal Women - Individualisation of Oestrogen Therapy
Acronym: OPTIMISE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Chelsea and Westminster NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013MM002B; 2013-002094-22 (EudraCT Number)
Record Dates: First submitted 2013-12-20; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Venous Thrombosis; Insulin Resistance
MeSH Terms: conditions — Venous Thrombosis; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femoston Conti 0.5mg/2.5mg (Experimental): Ultra low dose, film-coated 17β-estradiol (as hemihydrate) 0.5mg & dydrogesterone 2.5 mg
  Once a day
  The duration is six months.
  Drug intervention: Estradiol&DydrogesteronevsOestradiol&Norethisterone acetate
  Interventions: Drug: Femoston Conti
- EVOREL® CONTI transdermal patches (Active Comparator): EVOREL CONTI is a transdermal self adhesive patch which is 0.1 mm in thickness and each patch releases 50mcg of oestradiol and 170mcg of norethisterone acetate over 24 hours .
  The Evorel Conti patch is cut in half and applied to the lower part of the body for 3.5 days (delivering approx 25mcg of oestradiol over 24 hours ) this is replaced every 3.5 days .
  The duration is six months.
  Drug intervention: Estradiol&DydrogesteronevsOestradiol&Norethisterone acetate
  Interventions: Drug: EVOREL® CONTI

INTERVENTIONS:
Drug: Femoston Conti — Ultra-low-dose oral E2/D [Oestradiol 17β 0.5mg/dydrogesterone 2.5 mg] oral Femoston Conti 0.5mg Estradiol&Dydrogesterone vs Oestradiol&Norethisterone acetate
  Other Names: Femoston Conti 0.5mg/2.5mg film-coated tablets versus
  Arms: Femoston Conti 0.5mg/2.5mg
Drug: EVOREL® CONTI — Trans-dermal Estradiol 25mcg/norethisterone acetate 85 mcg 1/2 an Evorel Conti patch
  Other Names: Evorel Conti transdermal patch 25 mcg transdermal dose
  Arms: EVOREL® CONTI transdermal patches

SUMMARY:
Ultra-low-dose oral E2/D will have more beneficial effects than trans-dermal HRT on lipids and insulin resistance in postmenopausal women, whilst adverse effects on coagulation will be avoided.

DETAILED DESCRIPTION:
Following screening for eligibility, women will be studied at baseline and then randomized to one of two groups:

Group A administered Femoston Conti - oral oestradiol 17β 0.5 mg/dydrogesterone 2.5 mg daily for the duration of the treatment phase (24 weeks)

Group B administered ½ Evorel Conti patches - trans-dermal Estradiol 25 mcg/norethisterone acetate 85 mcg (½ Evorel Conti patches) daily for the duration of the treatment phase (24 weeks).

Studies will be repeated after 6 months of therapy at the follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and postmenopausal woman who have had a normal ultrasound result
* Aged 40 - 60 years
* At least 1 year post last menstrual period (per participant report)
* BMI 18 - 32
* Normal mammogram within 2 years of study commencement
* Continue on any concomitant medications without any change during the study give informed consent

Exclusion Criteria:

* Estrogen or androgen therapy during preceding 3 months
* Use of hormone implants during the preceding 12 months
* Have received any medications which may interfere with the study (SSRI, antiandrogens,
* PDE5 inhibitors, DHEA, SERMS)
* Have a significant psychiatric disorder
* Have a history of breast or oestrogen dependent cancer
* Have diabetes, thrombo-embolic disorders (recent MI angina DVT varicose veins or recurrent DVT), cardiovascular disease, liver disease any condition affecting carbohydrate metabolism, uncontrolled hypertension and uncontrolled hyperlipidaemia
* Untreated endometrial hyperplasia
* Dubin-Johnson syndrome and Rotor syndrome
* Undiagnosed vaginal bleeding
* Women who have had a hysterectomy

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Thrombin Generation IU/DL | Six months

SECONDARY OUTCOMES:
triglycerides | 6 months
  mmol/L
HDL | 6 months
  mmol/L
Total cholesterol | 6 months
  mmol/L
LDL | 6 months
  mmol/L
D-Dimers | 6 months
  ng/ml
APC resistance | 6 months
  >2 or <2
fibrinogen | 6 months
  g/L
Factor V11 | 6 months
  U/ml
PAI-1 protein | 6 months
  nq/ml
fasting insulin | 6 months
  pmol/L
fasting glucose | 6 months
  mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: John Stevenson, MBBS, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Chelsea and Westminster NHS Foundation Trust, London
  - Royal Brompton and Harefield NHS Trust, London
  - Imperial College Healthcare NHS Trust, London